CLINICAL TRIAL: NCT01253473
Title: COPDGene Ancillary Proposal: Symbicort Intervention in "Airway Predominant
Brief Title: Symbicort in Airway Predominant Chronic Obstructive Pulmonary Disease (COPD)
Acronym: SACOPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Jewish Health (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYMB0012
Record Dates: First submitted 2010-11-16; First posted 2010-12-03 (Estimated); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Budesonide; Budesonide, Formoterol Fumarate Drug Combination; Albuterol, Ipratropium Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ipratropium/albuterol (Active Comparator): 1 puff 4 times daily
  Interventions: Drug: Ipratropium/albuterol
- Budesonide (Experimental): budesonide 180 ug 2 puffs 4 times daily + ipratropium/albuterol 1 puffs four times daily
  Interventions: Drug: Budesonide; Drug: Ipratropium/albuterol
- budesonide/formoterol (Experimental): budesonide/formoterol 160/4.5 ug 2 puffs 4 times daily + ipratropium/albuterol 1 puffs four times daily
  Interventions: Drug: budesonide/formoterol; Drug: Ipratropium/albuterol

INTERVENTIONS:
Drug: Budesonide — Inhaled budesonide twice daily plus inhaled ipratropium/albuterol combination four times daily and every 4 hours as needed
  Other Names: Pulmicort Flexhaler®
  Arms: Budesonide
Drug: budesonide/formoterol — Inhaled budesonide/formoterol (160/4.5 mcg Symbicort®) 2 puffs twice daily plus inhaled ipratropium/albuterol (Combivent®) 1 puff four times daily
  Other Names: Symbicort®
  Arms: budesonide/formoterol
Drug: Ipratropium/albuterol — Inhaled ipratropium/albuterol combination 2 puffs four times daily
  Other Names: Combivent®

SUMMARY:
The main objective of the study is to see if using anti-inflammatory to patients with airway disease chronic obstructive pulmonary disease (COPD) phenotype will be more effective than using these treatments in patients with loss of lung tissue. Symbicort plus ipratropium/albuterol will be used for 12 weeks in an open-label study in subjects with airway predominant COPD.

DETAILED DESCRIPTION:
Subjects from the COPDGene study who have airway-predominant COPD on chest CT scan will be enrolled; a total of 40 subjects is planned.

Subjects will all have background ipratropium-albuterol administered four times daily. Subjects will be randomized to receive budesonide (180 ug twice daily) or formoterol-budesonide (160/4.5 ug twice daily) for 12 weeks.

The main objective is to explore novel outcomes: blood biomarkers and chest CT scan. Outcomes include lung function, walk distance, respiratory disease-specific health status, and expiratory chest CT scan gas trapping as an exploratory outcome.

The primary outcome measure will be FEV1 pre-bronchodilator 12 hours after the last dose of study medication at the end of 12 weeks of treatment. FEV1 will be measured in the morning 6 hours after the last dose of ipratropium/albuterol and 12 hours after the last dose of budesonide and budesonide/formoterol

ELIGIBILITY:
Inclusion Criteria:

1. COPD GOLD Stage 2 and 3 (post-bronchodilator FEV1 35-80% predicted and FEV1/FVC <0.7 at the time of enrollment in COPDGene) by spirometry.
2. Less than 15% of the lung <-950 Hounsfield Units on COPDGene high-resolution inspiratoryChest CT scan (i.e. no evidence of significant emphysema)
3. Greater than 10% gas trapping on COPDGene expiratory CT scan (i.e. evidence of small airway disease).
4. No history of recent use (within the pat 8 weeks) of an inhaled or systemic corticosteroid.
5. Body weight <100 kg (low dose CT scans in subject with increased boyd weight can not be reliably analyzed).

Exclusion Criteria:

1. Exacerbation of COPD or other respiratory illness requiring antibiotics within the past 8 weeks.
2. Previous adverse reaction to inhaled steroids, long-acting beta agonists, or long-acting anticholinergic medications.
3. Symptomatic, untreated benign prostate hypertrophy.
4. Allergy to peanuts.
5. Glaucoma

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Forced expiratory volume in 1 second (FEV1) pre-bronchodilator | 12 weeks
  FEV1 will be measured in the morning 6 hours after the last dose of ipratropium/albuterol and 12 hours after the last dose budesonide and budesonide/formoterol

SECONDARY OUTCOMES:
Health Status | 12 weeks
  Administer St. George's Respiratory Questionnaire at randomization and 12 weeks.
Dyspnea | 12 weeks
  Evaluated by the Modified Medical Research Council Dyspnea Scale at randomization and week 12.
Six minute walk distance | 12 weeks
  Evaluate six minute walk distance at randomization and 12 weeks
Forced vital capacity (FVC) pre-bronchodilator | 12 weeks
Post-bronchodilator FEV1 | 12 weeks
Patient-reported exacerbations | 12 weeks
Patient reported adverse events | 12 weeks
Post-bronchodilator FVC | 12 weeks
CT scan gas trapping | Before and 12 weeks after randomization

CONTACTS AND LOCATIONS:
Overall Officials: James D Crapo, MD, Principal Investigator — National Jewish Health; Edwin K Silverman, MD, PhD, Principal Investigator — Brigham and Women's Hospital; Barry J Make, MD, Principal Investigator — National Jewish Health
Locations (7):
- United States (7):
  - University of Alabama Birmingham Medical Center, Birmingham, Alabama
  - Harbor UCLA Medical Center, Torrance, California
  - National Jewish Health, Denver, Colorado
  - University of Iowa, Iowa City, Iowa
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Reliant Medical Group, Worcester, Massachusetts
  - Temple University Medical Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No